CLINICAL TRIAL: NCT02456272
Title: Hearing Aid Versus Surgical Rehabilitation as Treatment of Otosclerosis: Pilot Study
Acronym: PARCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/14/7312; 2014-A01764-43 (Other: ID-RCB)
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2018-05

CONDITIONS: Otosclerosis
Keywords: Otosclerosis; Surgical treatment; Hearing aids
MeSH Terms: conditions — Otosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- External hearing aid & Otosclerosis surgery (Experimental): Trying an hearing aid for at least two months and then undergo otosclerosis surgery
  Interventions: Device: External hearing aid; Procedure: Otosclerosis surgery

INTERVENTIONS:
Device: External hearing aid — The external hearing aid (monaural) with an auditory prosthesis contour type, brand PHONAK type Bolero Q70 will be provided to the patients during a minimum of 2 months.For reasons of standardization and comparability of results, only one type of prosthesis (medium-high range) will be provided. The settings will be performed by audiologists of ENT service during the inclusion visit.
Procedure: Otosclerosis surgery — Surgical restoration of the columellar effect consists of the intraoperative verification of the stapedo-vestibular ankylosis which provides diagnostic. Then a stapedotomy (laser or Ototool°) is performed and partial ossicular prosthesis s inserted between stapedotomy and the long process of the incus.

SUMMARY:
This is a French pilot study in the Toulouse University Hospital that will include a minimum of 30 patients with proven unilateral or asymmetric otosclerosis. Each one will receive a hearing aid for a minimum of 2 months and then undergo otosclerosis surgery.

DETAILED DESCRIPTION:
Otosclerosis is the main cause of acquired hearing loss in young to middle aged Caucasian population. Social, personal and medico-economic impacts triggered by this affection make it a major public health matter. Historically, the surgical treatment of otosclerosis has always been considered one of the best indications of otologic surgery. The external hearing aid was then an alternative to surgery considered as a more restrictive and less effective management of otosclerosis. With the recent technological developments of hearing aids, comparing these two treatments otosclerosis should be studied. The absence of scientific data from the literature concerning this subject justifies this study which purpose is to describe the evolution of the quality of life and hearing performance of a same patient after taking over by these two approaches.

This is a French pilot study in the Toulouse University Hospital that will include a minimum of 30 patients with proven unilateral or asymmetric otosclerosis. Each one will receive a hearing aid for a minimum of 2 months and then undergo otosclerosis surgery.

The primary outcome will be based on a study of the quality of life (score of 0-100 to quality of life validated questionnaire Glasgow Health Status Inventory (GHSI)). The questionnaire will be given to the patient at the pre-enrollment visit, after a period of two months of external hearing aid trying and 2 months after the surgery. Secondary outcomes will be studied: simple hearing performance (voice and tone audiogram), complex hearing performance (speech audiogram in noise recognition stamp), specific questionnaires for hearing (SSQ), for hearing aids (APHAB, GBI equipment), for tinnitus if present (THI and VAS discomfort / intensity) or for surgical treatment (surgery GBI). Data about treatment's side effects and the number of potential patients refusing surgery after testing the hearing aid will also be collected.

ELIGIBILITY:
Inclusion Criteria:

Nosological criteria:

* Unilateral or bilateral asymmetric otosclerosis
* Conductive hearing loss of at least 30 dB with an average loss Rinne means greater than or equal to 20 dB (on frequencies 0.5, 1, 2, 4 kHz)
* Normal tympanum
* Temporal bones CT-scan showing radiologic signs of otosclerosis

Related to treatment criteria:

• No previous treatment for the otosclerosis

Exclusion Criteria:

Disease's related criteria:

* Far advanced otosclerosis defined as less than 95dB air conduction at all frequencies or lower bone conduction 55dB on at least one frequency
* Cochlear otosclerosis objectified on the temporal bones Ct-scan
* Others clinical or radiological diagnostics: cholesteatoma, tympanic membrane perforation, geyser's syndrome, ossicular dislocation, ossicular malformation, tympanosclerosis.

Associated pathologies: tympanic retraction, effects of chronic otitis, tubal dysfunction.

Criteria about proposed treatments:

* Anesthesia contraindications
* Operative contraindication: clotting disorders, tympanum retraction and tubal dysfunction, geyser's syndrome, single ear, patient refusal.

Criteria relative to study's explorations: Language barrier (questionnaires, tests), cognitive disorders.

Criteria relating to previous treatment: Previous hearing aid or surgery Administrative criteria: Patients minors, incapable adults, adults under guardianship, incapable of giving consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Evolution of the quality of life (scored by GHSI) | 4th Month
  The primary outcome is to describe the evolution of the quality of life (scored by the Glasgow Health Status Inventory (GHSI)) during the hearing rehabilitation of otosclerosis frst with an external monaural hearing aid (support for at least 2 months), followed by a surgical treatment.

SECONDARY OUTCOMES:
Evolution of the quality of life (scored by SSQ) | Change and evolution at different time points: baseline, 2-month intervention, 2-month after surgery
  Secondary outcomes will be to describe the evolution of the quality of life by specific questionnaires (SSQ APHAB, GBI), the evolution of simple and complex audiometric testing in both managements of otosclerosis. Adverse reactions reported are also analyzed as well as the number of patients refusing surgery after trying hearing aid rehabilitation.
Evolution of the quality of life (scored by APHAB) | Change and evolution at different time points: baseline, 2-month intervention, 2-month after surgery
  Secondary outcomes will be to describe the evolution of the quality of life by specific questionnaires (SSQ APHAB, GBI), the evolution of simple and complex audiometric testing in both managements of otosclerosis. Adverse reactions reported are also analyzed as well as the number of patients refusing surgery after trying hearing aid rehabilitation.
Evolution of the quality of life (scored by GBI) | Change and evolution at different time points: baseline, 2-month intervention, 2-month after surgery
  Secondary outcomes will be to describe the evolution of the quality of life by specific questionnaires (SSQ APHAB, GBI), the evolution of simple and complex audiometric testing in both managements of otosclerosis. Adverse reactions reported are also analyzed as well as the number of patients refusing surgery after trying hearing aid rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu MARX, MD, Principal Investigator — Toulouse University Hospital (CHU Toulouse)
Locations (1):
- Toulouse University Hospital (CHU de Toulouse), Toulouse, France

REFERENCES:
- [Result] Molinier CE, Gallois Y, Deguine O, Iversenc G, Vales O, Taoui S, Lepage B, Fraysse B, Marx M. Stapedotomy Versus Hearing Aids in the Management of Conductive Hearing Loss Caused by Otosclerosis: A Prospective Comparative Study. Otol Neurotol. 2022 Aug 1;43(7):773-780. doi: 10.1097/MAO.0000000000003585. PMID 35878633